CLINICAL TRIAL: NCT04314284
Title: Implementing a Patient-Centered Intervention to Reduce Cancer Patients' Financial Toxicity
Brief Title: Patient-Centered Intervention to Reduce Cancer Patients' Financial Toxicity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 202003033; 1P50CA244431-01 (NIH)
Record Dates: First submitted 2020-03-16; First posted 2020-03-19 (Actual); Results first posted 2022-06-13 (Actual); Last update posted 2023-05-09 (Actual); Status verified 2023-05

CONDITIONS: Gynecologic Cancer; Colorectal Cancer; Lung Cancer
MeSH Terms: conditions — Colorectal Neoplasms; Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Historical Control Survey (Other): -The investigators will conduct a historic control survey of 80-100 recently diagnosed gynecologic, colorectal, and lung cancer patients. They can complete the survey in-person, over the phone, or online. The survey will take approximately 15 minutes to complete. It will ask about their knowledge of health insurance and confidence communicating about care costs.
  Interventions: Other: Historical control survey
- I Can PIC (Experimental): -Approximately 80-100 participants will use I Can PIC. This will take approximately 10-15 minutes. After their next appointment with their provider, they will complete a brief survey about their knowledge of health insurance and confidence communicating about care costs. This will take about 10 mins. Patient participants who choose to complete the study in person may view I Can PIC on a tablet provided in the clinic or at the office. Then after their appointment, they can complete the survey on a tablet provided in the clinic or at the office. If they choose to complete it over the phone, the investigators will email them the link to I Can PIC and then call them when it is time to complete the survey. If they wish to complete it online, the investigators will email them the link to I Can PIC, and then the survey after their appointment. After 3-6 months, participants will receive a 5-10 minute follow-up survey which they can complete in-person, online, or over the phone.
  Interventions: Behavioral: I Can PIC; Other: Post-intervention survey (I Can PIC participants); Other: Follow-Up survey (I Can PIC participants)

INTERVENTIONS:
Behavioral: I Can PIC — -Online decision tool that explains health insurance terms and health insurance terms, provides tips on lowering health care costs, advises patient to discuss costs with provider and insurance, and provides financial resources for patient.
  Arms: I Can PIC
Other: Historical control survey — -31 questions including overall experience with cancer care provider, previous discussions with care team regarding health care costs, preferences for discussing health care costs with physician, confidence level on discussing health care costs with physician, feelings about current financial situation, delays or avoidance of medical care in the past 12 months, confidence in health care choices and health insurance choices, current health conditions, and demographic data.
  Arms: Historical Control Survey
Other: Post-intervention survey (I Can PIC participants) — -31 questions including overall experience with cancer care provider, previous discussions with care team regarding health care costs, preferences for discussing health care costs with physician, confidence level on discussing health care costs with physician, feelings about current financial situation, delays or avoidance of medical care in the past 12 months, confidence in health care choices and health insurance choices, current health conditions, and demographic data.
  Arms: I Can PIC
Other: Follow-Up survey (I Can PIC participants) — -19 questions including overall experience with cancer care provider, discussion with care team regarding health care costs, preferences for discussing health care costs with physician, confidence level on discussing health care costs with physician, feelings about current financial situation, delays or avoidance of medical care in the past 12 months, and confidence in health care choices and health insurance choices.
  Arms: I Can PIC

SUMMARY:
The purpose of this study is to incorporate feedback from cancer patients and providers to adapt, implement, and test an intervention. The intervention aims to prompt screening for financial distress, facilitate discussions about care costs with cancer patients, support health insurance selection, and ultimately reduce cancer patients' financial toxicity associated with cancer care.

ELIGIBILITY:
Eligibility criteria for I Can Pic Arm only:

Inclusion Criteria:

* 18 years of age or older
* Must have been diagnosed with colorectal cancer, lung cancer, or gynecologic cancer < 5 months ago and be patients of one of the 15 providers
* This cancer diagnosis must be the first and primary diagnosis

Exclusion Criteria:

* Not able to read and understand English
* Cannot give informed consent due to cognitive or emotional barriers

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2020-05-26 (Actual); Primary Completion 2021-08-27 (Actual); Study Completion 2021-11-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mary Politi, Ph.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Historical Control Survey | I Can PIC
Started | 69 | 81
Completed | 65 | 68
Not Completed | 4 | 13
Not completed — Withdrawal by Subject | 4 | 7
Not completed — Consented but did not complete survey | 0 | 6

BASELINE CHARACTERISTICS:
Population: 3 participants who withdrew in the Historical Control Survey arm still provided their demographic data before withdrawing from the study and the demographic data is included. 1 participant in the I Can PIC arm did not provide their age which is why the number of participants for age, continuous is 67 and the total for age is 135.
Groups:
- Total: Total of all reporting groups
Arm/Group | Historical Control Survey | I Can PIC | Total
Number analyzed (Participants) | 68 | 68 | 136
Age, Continuous [Median (Full Range); unit: years] — Population: One participant in the I Can PIC arm did not provide their age.
  years
    number analyzed (Participants) | 68 | 67 | 135
    (all) | 61.5 [30 to 87] | 60 [27 to 84] | 61 [27 to 84]
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 40 | 43 | 83
  Male | 25 | 25 | 50
  Unknown | 3 | 0 | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 64 | 68 | 132
  Unknown or Not Reported | 3 | 0 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 3 | 7
  White | 58 | 65 | 123
  More than one race | 2 | 0 | 2
  Unknown or Not Reported | 3 | 0 | 3
Region of Enrollment [Number; unit: participants]
  United States | 68 | 68 | 136

OUTCOME MEASURES:

1. Primary Outcome: Difference in Health Insurance Knowledge Between Historical Control Arm and I Can PIC Arm
Description: * Health insurance knowledge will be collected on the historical control survey and the I Can PIC post-intervention survey
  * Score from 0% (worst) to 100% (best). Higher scores indicate greater health insurance knowledge
Time Frame: Completion of survey (estimated to be approximately 1-14 days after enrollment)
Population: 3 participants in the Historical Control Survey arm did not complete the survey.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Historical Control Survey | I Can PIC
Number analyzed (Participants) | 65 | 68
score on a scale | 72.45 (18.77) | 77.02 (19.03)
Statistical Analysis 1: Comparison: Historical Control Survey vs I Can PIC; Test type: Superiority; p = 0.15, Kruskal-Wallis

2. Primary Outcome: Difference in Health Insurance Literacy Between Historical Control Arm and I Can PIC Arm
Description: * Health insurance literacy will be collected on the historical control survey and the I Can PIC post-intervention survey
  * Score from 12 (worst) to 48 (best). Higher scores indicate greater health insurance literacy
Time Frame: Completion of survey (estimated to be approximately 1-14 days after enrollment)
Population: 3 participants in the Historical Control Survey arm did not complete the survey.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Historical Control Survey | I Can PIC
Number analyzed (Participants) | 65 | 68
score on a scale | 33.03 (8.56) | 34.71 (7.65)
Statistical Analysis 1: Comparison: Historical Control Survey vs I Can PIC; Test type: Superiority; p = 0.35, Kruskal-Wallis

3. Primary Outcome: Difference in the Number of Clinicians That Discussed Health Care Cost Topics With Participants Between the Historical Control Arm and I Can PIC Arm
Description: * Information regarding clinicians who discussed health care costs will be collected on the historical control survey and the I Can PIC post-intervention survey
  * Score either no (did not discuss health care costs with clinician) or yes (discussed one more cost-related topics with clinicians)
  * Also score the number of cost-related topics discussed, if yes
Time Frame: Completion of survey (estimated to be approximately 1-14 days after enrollment)
Measure: Count of Participants; unit: Participants
Arm/Group | Historical Control Survey | I Can PIC
Number analyzed (Participants) | 68 | 68
Participants | 46 | 39
Statistical Analysis 1: Comparison: Historical Control Survey vs I Can PIC; Test type: Superiority; p = 0.22, Chi-squared

4. Primary Outcome: Difference in the Number of Cost-related Topics Discussed With Participants Between the Historical Control Arm and I Can PIC Arm
Description: -Information regarding clinicians who discussed health care costs will be collected on the historical control survey and the I Can PIC post-intervention survey
Time Frame: Completion of survey (estimated to be approximately 1-14 days after enrollment)
Measure: Number; unit: cost-related topics discussed
Arm/Group | Historical Control Survey | I Can PIC
Number analyzed (Participants) | 68 | 68
cost-related topics discussed
  Insurance eligibility or coverage | 32 | 33
  Time off work during treatment or recovery | 16 | 15
  Cost of drugs to treat cancer | 9 | 11
  Costs of getting to and from visits | 8 | 1
  Costs of specific tests, visits, or equipment | 7 | 5
  Cost of over-the-counter drugs | 3 | 6
  Comparing costs of options to help choose care | 3 | 0
  Cost of day-to-day living | 2 | 2
  Other | 1 | 2

5. Primary Outcome: Difference in the Number of Clinicians That Discussed Health Care Cost Strategies Between the Historical Control Arm and I Can PIC Arm
Description: as for outcome 4
Time Frame: Completion of survey (estimated to be approximately 1-14 days after enrollment)
Measure: Count of Participants; unit: Participants
Arm/Group | Historical Control Survey | I Can PIC
Number analyzed (Participants) | 68 | 68
Participants | 32 | 33

6. Primary Outcome: Difference in the Number of Cost Strategies Discussed Between the Historical Control Arm and I Can PIC Arm
Description: as for outcome 4
Time Frame: Completion of survey (estimated to be approximately 1-14 days after enrollment)
Measure: Number; unit: cost strategies discussed
Arm/Group | Historical Control Survey | I Can PIC
Number analyzed (Participants) | 68 | 68
cost strategies discussed
  Changing logistics of care | 21 | 18
  Change the dose (amount) of treatment | 7 | 8
  Choosing a generic drug instead of a brand name drug | 6 | 8
  Setting up a payment plan | 2 | 12
  Copay assistance, coupons, or rebates for drugs | 2 | 6
  Referring to hospital billing office | 8 | 5
  Stopping or pausing some treatments | 4 | 3
  Suggesting a community agency or charity | 2 | 2
  Suggesting a free drug program | 1 | 0
  Suggesting talking to human resources | 1 | 0
  Choosing a lower cost procedure or scan | 0 | 0
  Suggesting government assistance | 0 | 0
  Other | 4 | 1

7. Primary Outcome: Difference in Confidence Communicating About Health Care Costs With Physician Between Historical Control Arm and I Can PIC Arm
Description: * Confidence communicating about health care costs will be collected on the historical control survey and the I Can PIC post-intervention survey
  * Score from 4 (worst) to 16 (best). Higher scores indicate greater confidence communicating about care costs
Time Frame: Completion of survey (estimated to be approximately 1-14 days after enrollment)
Population: 4 participants in the Historical Control Survey arm did not complete the survey.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Historical Control Survey | I Can PIC
Number analyzed (Participants) | 64 | 68
score on a scale | 13.59 (2.92) | 13.81 (2.75)
Statistical Analysis 1: Comparison: Historical Control Survey vs I Can PIC; Test type: Superiority; p = 0.65, Kruskal-Wallis

8. Primary Outcome: Difference in Financial Toxicity Between Historical Control Arm and I Can PIC Arm
Description: * Financial toxicity will be collected on the historical control survey and the I Can PIC post-intervention survey
  * Score from 0 (best) to 44 (worst). Higher scores indicate greater financial toxicity
Time Frame: Completion of survey (estimated to be Day 1 for historical control participants and estimated to be Day 14 for I Can PIC participants)
Population: 3 participants in the Historical Control Survey arm did not complete the survey
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Historical Control Survey | I Can PIC
Number analyzed (Participants) | 65 | 68
score on a scale | 17.71 (11.20) | 16.06 (9.83)
Statistical Analysis 1: Comparison: Historical Control Survey vs I Can PIC; Test type: Superiority; p = 0.52, Kruskal-Wallis

9. Primary Outcome: Difference in Number of Clinicians Who Referred Patients to Resources to Discuss Costs
Description: * Information regarding clinicians who discussed health care costs will be collected on the historical control survey and the I Can PIC post-intervention survey
  * Score either no (did not refer to resources) or yes (referred to resources)
  * Also score the number of cost-related topics discussed, if yes
Time Frame: Completion of survey (estimated to be approximately 1-14 days after enrollment)]
Measure: Count of Participants; unit: Participants
Arm/Group | Historical Control Survey | I Can PIC
Number analyzed (Participants) | 68 | 68
Participants | 11 | 14
Statistical Analysis 1: Comparison: Historical Control Survey vs I Can PIC; Test type: Superiority; p = 0.51, Chi-squared

10. Secondary Outcome: Health Insurance Knowledge Sustained Over Time (I Can PIC Arm)
Description: * Sustained Health insurance knowledge will be collected on the post-intervention survey and the 3-6 month follow-up survey
  * Score from 0% (worst) to 100% (best). Higher scores indicate greater health insurance knowledge
Time Frame: Change from post-intervention survey to 3-6 month follow-up survey (estimated to be a total of 6 months)
Population: Only participants enrolled in the I Can PIC Arm were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Historical Control Survey | I Can PIC
Number analyzed (Participants) | 0 | 68
score on a scale
  Post-intervention survey |  | 77.02 (19.03)
  3-6 month follow-up survey: number analyzed (Participants) | 0 | 63
  3-6 month follow-up survey |  | 75.6 (20.01)

11. Secondary Outcome: Health Insurance Literacy Sustained Over Time (I Can PIC Arm)
Description: * Sustained Health insurance literacy will be collected on the post-intervention survey and the 3-6 month follow-up survey
  * Score from 12 (worst) to 48 (best). Higher scores indicate greater health insurance literacy
Time Frame: Change from post-intervention survey to 3-6 month follow-up survey (estimated to be a total of 6 months)
Population: Only participants enrolled in the I Can PIC Arm were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Historical Control Survey | I Can PIC
Number analyzed (Participants) | 0 | 68
score on a scale
  Post-intervention survey |  | 34.71 (7.65)
  3-6 month follow-up survey: number analyzed (Participants) | 0 | 65
  3-6 month follow-up survey |  | 35.74 (8.39)

12. Secondary Outcome: Confidence Communicating About Health Care Costs With Physician (I Can PIC Arm)
Description: * Confidence communicating about health care costs will be collected on the post-intervention survey and the 3-6 month follow-up survey
  * Score from 4 (worst) to 16 (best). Higher scores indicate greater confidence communicating about care costs
Time Frame: Change from post-intervention survey to 3-6 month follow-up survey (estimated to be a total of 6 months)
Population: Only participants enrolled in the I Can PIC Arm were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Historical Control Survey | I Can PIC
Number analyzed (Participants) | 0 | 68
score on a scale
  Post-intervention survey |  | 13.81 (2.75)
  3-6 month follow-up survey: number analyzed (Participants) | 0 | 63
  3-6 month follow-up survey |  | 14.24 (2.47)
Statistical Analysis 1: Comparison: Historical Control Survey vs I Can PIC; Test type: Other — 2-sided; p = 0.71, t-test, 2 sided

13. Secondary Outcome: Sustained Financial Toxicity (I Can PIC Arm)
Description: * Sustained Financial toxicity will be collected on the post-intervention survey and the 3-6 month follow-up survey
  * Score from 0 (best) to 44 (worst). Higher scores indicate greater financial toxicity
Time Frame: Change from post-intervention survey to 3-6 month follow-up survey (estimated to be a total of 6 months)
Population: Only participants enrolled in the I Can PIC Arm were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Historical Control Survey | I Can PIC
Number analyzed (Participants) | 0 | 68
score on a scale
  Post-intervention survey |  | 16.06 (9.83)
  3-6 month follow-up survey: number analyzed (Participants) | 0 | 63
  3-6 month follow-up survey |  | 14.17 (10.72)
Statistical Analysis 1: Comparison: I Can PIC; Test type: Other — 2-sided; p = 0.12, t-test, 2 sided

14. Other Pre Specified Outcome: Delayed or Forgone Care Due to Costs (I Can PIC Arm)
Description: * Delayed or forgone care due to costs will be collected on the post-intervention survey and the 3-6 month follow-up survey
  * Score from 0 (best) to 8 (worst). Higher scores indicate more frequent delayed and forgone care due to costs
Time Frame: Change from post-intervention survey to 3-6 month follow-up survey (estimated to be a total of 6 months)
Population: Only participants enrolled in the I Can PIC Arm were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Historical Control Survey | I Can PIC
Number analyzed (Participants) | 0 | 68
score on a scale
  Post-intervention survey |  | 2.33 (1.58)
  3-6 month follow-up survey: number analyzed (Participants) | 0 | 63
  3-6 month follow-up survey |  | 2.38 (1.50)

15. Other Pre Specified Outcome: Delayed or Forgone Care Due to Costs (Historical Control Arm and I Can PIC Arm)
Description: * Delayed or forgone care due to costs will be collected on the historical control survey and the I Can PIC post-intervention survey
  * Score from 0 (best) to 8 (worst). Higher scores indicate more frequent delayed and forgone care due to costs
Time Frame: Completion of survey (estimated to be approximately 1-14 days after enrollment)
Population: 3 participants in the Historical Control Survey arm did not complete the survey.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Historical Control Survey | I Can PIC
Number analyzed (Participants) | 65 | 68
score on a scale | 2.67 (1.61) | 2.33 (1.58)
Statistical Analysis 1: Comparison: Historical Control Survey vs I Can PIC; Test type: Superiority; p = 0.66, Kruskal-Wallis

ADVERSE EVENTS:
Time Frame: From start of study through completion of study (estimated to be 3-6 months).
Arm/Group | Historical Control Survey | I Can PIC
All-Cause Mortality (participants affected / at risk) | 7/68 | 2/68
Serious Adverse Events (participants affected / at risk) | 0/68 | 0/68
Other Adverse Events (participants affected / at risk) | 0/68 | 0/68

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-09-07): https://cdn.clinicaltrials.gov/large-docs/84/NCT04314284/Prot_SAP_000.pdf
  • Informed Consent Form (2020-10-27): https://cdn.clinicaltrials.gov/large-docs/84/NCT04314284/ICF_001.pdf